CLINICAL TRIAL: NCT06835088
Title: Cryopreservation Of Ovarian Tissue: Assessment Of Reimplantation Rate And Effects On Ovarian Function
Brief Title: Cryopreservation of Ovarian Tissue: Reimplantation Rate and Effects on Ovarian Function
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CRIO-2021
Record Dates: First submitted 2024-11-28; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Cryopreservation
Keywords: cryopreservation; ovarian tissue; ovarian function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature ovarian failure (POI) is a clinical syndrome defined by the loss of ovarian activity before age 40. POI is characterized by amenorrhea or oligomenorrhea with elevated gonadotropins, low estradiol and serious consequences on fertility.

The prevalence of POI in the general population is about 1%. In recent years, the incidence of iatrogenic POI in cancer women is increasing: 4% of patients of fertile age are diagnosed with neoplasms and gonadal treatments that can sterilize them, such as chemotherapy and radiotherapy. Preserving fertility is a key objective for many cancer patients.

Before gonadotoxic treatments, patients in the post-pubertal age with future desire for pregnancy may opt for two main methods of preservation of fertility (FP): egg cryopreservation (OC) after ovarian stimulation and cryopreservation of ovarian tissue (OTC). An important limitation of the latter technique is the reduced number of patients who return to use the cryopreserved material, leading to a negative impact on the evaluation of the effectiveness of the procedure. The best way to maximise the effectiveness of the procedure in clinical and economic terms would be to increase the number of patients who continue the cryopreservation path by completing it with subsequent reimplantation. It would also be useful to improve the follow-up of these patients by evaluating their ovarian function over time, before and after the removal and reimplantation, through the study of bone metabolism, cardiovascular risk and psychological function in these women.

DETAILED DESCRIPTION:
Premature ovarian failure (POI) is a clinical syndrome defined by the loss of ovarian activity before age 40. POI is characterized by amenorrhea or oligomenorrhea with elevated gonadotropins, low estradiol and serious consequences on fertility. The prevalence of POI in the general population is about 1%. In recent years, the incidence of iatrogenic POI in cancer women is increasing: 4% of patients of fertile age are diagnosed with neoplasms and gonadal treatments that can sterilize them, such as chemotherapy and radiotherapy. Preserving fertility is a key objective for many cancer patients. The American Society of Clinical Oncology (ASCO) says that healthcare professionals who care for cancer patients should address infertility as soon as possible before starting treatment. In addition, the demand for fertility preservation for non-oncology diseases as well as personal reasons has increased significantly, and meeting this demand is a major challenge.

Before gonadotoxic treatments, patients in the post-pubertal age with future desire for pregnancy may opt for two main methods of preservation of fertility (FP): egg cryopreservation (OC) after ovarian stimulation and cryopreservation of ovarian tissue (OTC). The OC has been proven to be a reproducible, safe and effective technique for several years. However, it has some important limitations: OC may delay the start of treatment for cancer; in some specific types of cancer, ovarian stimulation should be avoided; the technique cannot be performed in prepubertal patients.

In these cases, OTC, a technique which has emerged from its experimental phase, now safe and with an increasing number of successes, is considered as the unique option for FP. Also, unlike OC, OTC allows the induction of puberty in prepubertal patients, restoration of ovarian hormonal function for 3-7 years, until the graft is active, and may be renewed by subsequent reimplantation of orthotopic or heterotropic tissue.

An important limitation of this technique is the reduced number of patients who return to use the cryopreserved material, which has a negative impact on the evaluation of the effectiveness of the procedure. Several causes in the period between ovarian sampling and transplantation may justify this low rate, including: i) loss of desire for pregnancy; ii) recurrence of cancer; iii) death of the patient; iv) financial reasons; ) fear of cancer recurrence due to contamination of ovarian sampling; vi) occurrence of spontaneous pregnancies; vii) absence of current partner.

The best way to maximise the effectiveness of the procedure in clinical and economic terms would be to increase the number of patients who continue the cryopreservation path by completing it with subsequent reimplantation. It would also be useful to improve the follow-up of these patients by evaluating their ovarian function over time, before and after the removal and reimplantation, through the study of bone metabolism, cardiovascular risk and psychological function in these women.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-55 years
* Suffering from diseases that require gonadotropic treatments
* Have been subjected to sampling and cryopreservation of ovarian tissue at the Operative Unit of Gynecology and Pathophysiology of Human Reproduction of the Sant'Orsola Polyclinic in Bologna
* Informed Consent Acquisition

Exclusion Criteria:

- Oncological pathology still active or relapse

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women aged between 13 and 55 years old suffering from oncological pathologies that require gonadotoxic treatments and who undergo prior to these treatments a collection of ovarian tissue for cryopreservation and possible subsequent orthotopic or heterotropic reimplantation in order to restore ovarian function and fertility
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Causes and factors that influence the low rate of reimplantation of ovarian tissue | At least 5 years after surgery at first follow-up
  Investigate the causes and factors that influence the low rate of reimplantation of ovarian tissue after the phase of collection and cryopreservation
Early ovarian failure | At least 5 years after surgery at first follow-up
  Effects of early ovarian failure in this category of women, particularly in terms of bone metabolism (through Bone densitometry with a dual-energy x-ray absorptiometry, DEXA, Z-score. BMD:> -2.0 normal; ≤ -2.0:osteoporosi
Early ovarian failure | At least 5 years after surgery at first follow-up
  Effects of early ovarian failure in this category of women, particularly in terms of cardiovascular risk (through ACC/AHA Cardiovascular Risk Calculator, %: <5%: low risk; 5-7.4%: Borderline risk; 7.5-19.9%: intermediate risk; ≥20%: high risk)
Early ovarian failure | At least 5 years after surgery at first follow-up
  Effects of early ovarian failure in this category of women, particularly in terms of psychological function (through Short Form36 HealthSurvey (SF-36), score: 0-100
Early ovarian failure | At least 5 years after surgery at first follow-up
  Effects of early ovarian failure in this category of women, particularly in terms of Middlesex Hospital Questionnaire (MHQ), score: <23: normal; >= 23: abnormal
Early ovarian failure | At least 5 years after surgery at first follow-up
  Effects of early ovarian failure in this category of women, particularly in terms of psychological function through Beck's Depression Inventory, score: 0-63

CONTACTS AND LOCATIONS:
Overall Officials: Renato Seracchioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy